CLINICAL TRIAL: NCT06145724
Title: EnCoRe MoMS Aim 1: Develop and Implement a Community-informed Institutional Obstetric Sepsis Bundle
Brief Title: EnCoRe MoMS: Engaging Communities to Reduce Morbidity From Maternal Sepsis (Aim 1)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Northern Manhattan Perinatal Partnership (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dena Goffman, Ellen Jacobson Levine and Eugene Jacobson Professor of Women's Health (in Obstetrics and Gynecology), Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAU3697 - Aim 1; 1UG3HD111247 (NIH)
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Maternal Sepsis; Infections
Keywords: Post Partum Period; Pregnancy; Maternal Health; Electronic Health Record
MeSH Terms: conditions — Pregnancy Complications, Infectious; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Admitted for Delivery (Comparing Pre vs Post-Implementation) (Experimental): Patients admitted for delivery at one of the partnering hospitals. EHR records from Columbia, Lincoln, Harlem, and Allen hospitals will be reviewed to evaluate process and outcome measures post-maternal sepsis bundle implementation. EHR data will be used from delivery hospitalizations.
  Interventions: Behavioral: Maternal Sepsis Safety Bundle

INTERVENTIONS:
Behavioral: Maternal Sepsis Safety Bundle — Maternal sepsis safety bundle implemented at Columbia, Lincoln, Harlem, and Allen hospitals.

SUMMARY:
Sepsis is the second leading cause of maternal death in the U.S. Labor and postpartum are particularly vulnerable risk periods. The goal of this multi-center, multidisciplinary study is to evaluate a maternal sepsis safety bundle.

DETAILED DESCRIPTION:
Maternal sepsis is the second leading cause of maternal death, major cause of morbidity, and preventable in most cases. Labor, birth, and postpartum are periods of increased sepsis risk. While American College of Obstetricians and Gynecologists (ACOG) and the Society for Maternal-Fetal Medicine (SMFM) recommend the implementation of safety bundles to prevent maternal mortality as the standard of care, there is limited evidence regarding effectiveness. EnCoRe MoMS will directly evaluate safety bundle performance for maternal sepsis. With extensive community partnerships and community organized leadership advisory board (CoLAB), EnCoRe MoMS: Engaging Communities to Reduce Morbidity from Maternal Sepsis will develop, implement, and evaluate a community-informed maternal sepsis bundle in 4 New York City (NYC) hospitals.

In Aim 1a: a robust community engagement and research infrastructures were established to design a comprehensive obstetric sepsis bundle that i) applies and optimizes standard evidence-based components of readiness, recognition, response, reporting, and respectful care ii) incorporates multidisciplinary obstetric provider training, and iii) integrates screening for unmet needs.

In Aim 1b, the investigators will assess participant outcomes pre- and post-maternal sepsis bundle implementation. Participants will be followed through their hospitalization until delivery hospitalization discharge or development of sepsis and readmissions pertinent to the study will be assessed. For the pre-implementation cohort, the investigators will use electronic health record (EHR) data from delivery hospitalizations to women from 2020-2022 from the four partner NYC hospitals compared to deliveries post-implementation (2025)during award period.

In the UH3 phase, the investigators will engage the community to implement the maternal sepsis care model, analyze results, and translate findings. Aim 1b. Implement the comprehensive obstetric sepsis bundle and evaluate its effectiveness using process and outcome measures Aim 1c. Define patterns in EHR of provider response to suspected sepsis, pre- vs post-bundle implementation; analyze associations between provider response variation and outcomes.

ELIGIBILITY:
Inclusion Criteria:

Birthing Person (EMR evaluation):

-Delivery hospitalizations and associated postpartum readmissions at the 4 hospital sites between 2020-2025

Exclusion Criteria:

Birthing Person (EMR evaluation)

-Delivery hospitalizations (and associated postpartum readmissions)to a hospital other than the 4 hospital sites or outside of 2020-2025 timeframe

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33183 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Diagnosed with Maternal Sepsis | Delivery Admission
  The number of patients diagnosed with maternal sepsis pre- and post- material sepsis bundle implementation. Sepsis as evaluated by the following scoring systems: Sepsis-2 (proven or suspected infection in combination with at least two systemic inflammatory response syndrome criteria); Sepsis-3 (organ dysfunction as defined by an acute change in total organ dysfunction score within 24 hours of suspected infection); and Center for Disease Control (CDC) Sepsis (presumed infection and organ dysfunction based on CDC criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Dena Goffman, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Columbia Unviersity Irving Medical Center, New York, New York
  - NewYork-Presbyterian Allen Hospital, New York, New York
  - NYC Health+Hospitals/Harlem, New York, New York
  - NYC Health + Hospitals/Lincoln, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No